CLINICAL TRIAL: NCT05679310
Title: Innovative Biotechnological Production of Antioxidant Products of Plant Origin From Microbial Factories, and Essential Oils From the Greek Flora, for the Creation of New Quality Health Products and Nutritional Supplements
Brief Title: Innovative Biotechnological Production of Antioxidant Products
Acronym: Antiox-Plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Patra Vezyraki, Professor, University of Ioannina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 82436
Record Dates: First submitted 2022-11-30; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Oxidative Stress; Inflammation; Body Weight; Homocystine; Metabolic Disorder
MeSH Terms: conditions — Inflammation; Body Weight; Metabolic Diseases | interventions — 3,4-dihydroxyphenylethanol; Oils, Volatile

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supplement (Experimental): The supplement capsules were given to 12 healthy subjects, aged 26-52, once a day for 8 weeks
  Interventions: Dietary Supplement: Hydroxytyrosol/Essential oils

INTERVENTIONS:
Dietary Supplement: Hydroxytyrosol/Essential oils — A dietary supplement containing 10 mg of hydroxytyrosol, synthesised using genetically modified Escherichia coli strains and equal amounts (8.33 μL) of essential oils from oregano vulgaris, sage officinalis and crithmum maritimum.

SUMMARY:
Several natural compounds have been explored as immune-boosting, antioxidant, and anti-inflammatory dietary supplements. Amongst them, hydroxytyrosol a natural antioxidant found in olive products, and endemic medicinal plants have attracted the scientific's community and industry's interest. The safety and biological activity of a standardised supplement containing 10 mg of hydroxytyrosol synthesized using genetically modified Escherichia coli strains and equal amounts (8.33 μL) of essential oils from oregano vulgaris, sage officinalis and crithmum maritimum in an open-label, single-arm, prospective clinical study were studied. The supplement capsules were given to 12 healthy subjects, aged 26-52, once a day for 8 weeks.

DETAILED DESCRIPTION:
The study was designed to evaluate the safety and biological activity of the supplement Antiox-Plus: one capsule/day, 15 minutes before their main meal which contained 10 mg of HT, synthesised using genetically modified Escherichia coli strains and equal amounts (8.33 μL) of essential oils from Origanum vulgare, Sage officinalis and Crithmum maritimum. The volunteers will consume the supplement for 8 weeks. A follow-up analysis will be performed one month after the end of the supplementation period (12 weeks from the initiation of the study). During this time, the participants will consume a placebo.

The volunteers are instructed to maintain their normal dietary habits. The following measurements will be taken: A) Dietary assessment at the beginning of the study (week 0), B) Body composition analysis at the beginning (week 0) and the end of the study (week 8), C) biochemical and laboratory analysis of plasma samples at week 0, 8 and 12.

The volunteers will record their food intake for 3 days (including one day of the weekend) and will fulfil a food frequency questionnaire. Analysis of their data will be done by a certified nutritionist. Nutritional assessment will be performed using the Evexis dietary software. The Tanita Dual Frequency Body Composition Monitor "Innerscan" will be employed to measure weight, muscle mass, muscle quality score, heart rate, body fat (%), physique rating, visceral fat, metabolic age, basal metabolic rate, bone mass, body water (%) and body mass index (BMI) in the morning. Physical activity will be assessed by the Greek version of the short International Physical Activity Questionnaire (IPAQ-short).

ELIGIBILITY:
Inclusion Criteria:

* age between 25 and 65 years
* the absence of any chronic health conditions
* adequate understanding of the study

Exclusion Criteria:

* the presence of any chronic health conditions (diabetes, hypertension, dyslipidemia)
* intake of nutritional supplements over the past 60 days
* heavy smokers (≥25 cigarettes/day)
* high alcohol use (men >14 drinks/week, women >7 drinks/week)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Homocysteine | Change from Baseline up to 12 weeks
  Homocysteine (μmol/L)
Fasting blood glucose | Change from Baseline up to 12 weeks
  Fasting blood glucose (md/dL)
oxLDL | Change from Baseline up to 12 weeks
  oxLDL (mU/mL)

SECONDARY OUTCOMES:
LDL-cholesterol | Change from Baseline up to 12 weeks
  LDL-cholesterol (mg/dL)
HDL-cholesterol | Change from Baseline up to 12 weeks
  HDL-cholesterol (mg/dL)
Glutathione | Change from Baseline up to 12 weeks
  Glutathione (mU/mL)
Catalase | Change from Baseline up to 12 weeks
  Catalase (units/mL)

OTHER OUTCOMES:
Total Antioxidant Capacity | Change from Baseline up to 12 weeks
  Total Antioxidant Capacity (mM a-tocopherol)
Malonaldehyde | Change from Baseline up to 12 weeks
  Malonaldehyde (μΜ)

CONTACTS AND LOCATIONS:
Overall Officials: Patra Vezyraki, PhD, Principal Investigator — University of Ioannina, School of Health Sciences, Department of Medicine, Laboratory of Physiology
Locations (1):
- University of Ioannina, Ioannina, Epirus, Greece